CLINICAL TRIAL: NCT04643821
Title: N-Acetylcysteine and Vitamin D in Infants With Hypoxic Ischemic Encephalopathy Treated With Hypothermia
Brief Title: NVD in Hypothermic HIE Neonates
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Dorothea D. Jenkins, Professor of Pediatrics, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 31254; 5F31NS108623-02 (NIH); FISPI14/0433 (Other Grant/Funding Number: Instituto Carlos III); 300118 (Other Grant/Funding Number: NIHR); P960743 (Other Grant/Funding Number: NIHR); EC11-246 (Other Grant/Funding Number: Spanish Ministry of Health, Social Services and Equality)
Record Dates: First submitted 2020-11-11; First posted 2020-11-25 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: HIE - Perinatal Hypoxic - Ischemic Encephalopathy
Keywords: oxidative stress; glutathione; pharmacokinetics
MeSH Terms: interventions — Acetylcysteine; Calcitriol

STUDY DESIGN:
Intervention Model Description: Open-label, escalating dose design
Who Masked: Outcomes Assessor
Masking Description: unaware of dose or timing of Magnetic resonance spectroscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- NAC 25mg/kg, calcitriol 0.05mcg/kg (Experimental): N-acetylcysteine 25mg/kg iv q 12h, calcitriol 0.05mcg/kg iv q 12h, for 10 days, starting within 6h of birth
  Interventions: Drug: N-acetylcysteine, NAC, and calcitriol
- NAC 25mg/kg, calcitriol 0.03mcg/kg (Experimental): N-acetylcysteine 25mg/kg iv q 12h, calcitriol 0.03mcg/kg iv q 24h, for 10 days, starting within 6h of birth
  Interventions: Drug: N-acetylcysteine, NAC, and calcitriol
- NAC 40mg/kg, calcitriol 0.03mcg/kg (Experimental): N-acetylcysteine 40mg/kg iv q 12h, calcitriol 0.03mcg/kg iv q 24h, for 10 days, starting within 6h of birth
  Interventions: Drug: N-acetylcysteine, NAC, and calcitriol

INTERVENTIONS:
Drug: N-acetylcysteine, NAC, and calcitriol — iv administration of antioxidant and active vitamin D
  Other Names: hypothermia

SUMMARY:
Neonatal hypoxic ischemic (HI) injury is an unpredictable neurologic injury with devastating, long term consequences for parents who are expecting a normal child. Hypothermia for 72 hr within 6 hrs of birth improves the combined outcome of death or severe disability, and hypothermia is now standard of care in tertiary centers throughout the world. However, approximately 50% of infants with hypoxic ischemic encephalopathy (HIE) treated with hypothermia still have adverse neurologic outcomes, due to ongoing neuroinflammation and oxidative stress in spite of hypothermia. Further, the majority of HIE infants are insufficient or deficient in a critical neurosteroid, 25(OH)vitamin D, which has been shown to adversely affect outcome after adult stroke. By adding vitamin D to N-acetylcysteine (NAC), an antioxidant, the investigators hypothesized that both drugs would increase glutathione (GSH) concentrations in critical brain areas, mitigate continuing oxidative stress after injury during hypothermia and after rewarming, and improve neurodevelopmental outcomes.

This is an open-label, non-randomized, escalating dose, pilot trial to evaluate the disposition and safety of NAC in combination with active vitamin D in neonates who present within 6 hrs of hypoxia ischemia/asphyxial event and received moderate hypothermia to 33 degrees C for 72 hours per routine protocol.

DETAILED DESCRIPTION:
N-acetylcysteine (NAC) is an FDA-approved drug that has been used in multiple conditions to mitigate oxidative stress. The study investigators' lab and others have shown that NAC provides neuroprotection either alone or in combination with hypothermia when given within 1-6 hrs of insult in animal models of HI injury. However, in neonatal rats subjected to severe hypoxic ischemic insult, NAC + hypothermia did not neuroprotect males as well as females. The study investigators and others determined that the majority of HIE infants are insufficient or deficient in 25(OH)vitamin D, a critical neurosteroid that also augments synthesis of an important antioxidant, glutathione. By adding active, low-dose 1,25-dihydoxy-Vitamin D3 to NAC (NVD), with a 1 hour delay after starting hypothermia, and repeated daily for 14 days in neonatal rat HI model, the study investigators significantly improved severity of brain injury over hypothermia alone in both sexes. Importantly, NVD also significantly improved functional outcomes of strength, sensorimotor and memory functioning 6 weeks after HI, even in male rats with the most severe brain pathology.

NAC and active vitamin D are FDA approved and are safe even in very sick newborns. In the study investigators' trial of NAC in maternal chorioamnionitis, comprehensive physiologic monitoring in preterm and term infants exposed to intrauterine inflammation demonstrated no significant differences in cerebral blood flow, oxygenation, or left ventricular function in infants treated with NAC or saline.

The primary objective of this study in human neonates after HIE birth treated with the standard hypothermia protocol, is to determine the unique pharmacokinetic (PK) parameters of NAC and vitamin D during hypothermia and after rewarming, verify the central nervous system (CNS) effect of NVD on the pharmacodynamic target, reduced glutathione, and determine the duration of CNS effect. The study investigators used low dose NAC (Acetadote, 25-40 mg/kg/dose) every 12 hours and Vitamin D3 (Calcitriol, 0.03 to 0.1microgram/kg) every 12-24 hours, infused IV for 10 days in a dose escalating study. The study investigators determined PK parameters and plasma oxidative stress markers during day 1 of life while hypothermic, and day 5 of life during normothermia (24-36 hours after rewarming). To establish effective dosing of NVD based directly on CNS effect, CNS metabolites were quantified with magnetic resonance spectroscopy (MRS) before and immediately after NVD dosing on DOL 5, infusing NVD during the routine MRI for HIE. In a subset of 10 infants the delayed effects of NVD on CNS metabolomics were determined by MRS between 2-6h after NVD dosing on DOL 5. Development was followed for >24months.

ELIGIBILITY:
Inclusion Criteria:

* Neonates > 34 weeks, > 2000 grams, within 6h of birth with moderate to severe HIE receiving therapeutic hypothermia

Exclusion Criteria:

* Evidence of a congenital CNS malformation if known prior to enrollment
* Evidence of neuromuscular disorder by family history
* More than 6 hours from birth or known insult
* Suspected genetic abnormality

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in pharmacokinetic half life of NAC | first week of life
  PK parameters of plasma half life around first dose on day of life 1 during hypothermia, and day of life 5 during normothermia
pharmacokinetic half life of calcitriol | first week of life
  PK parameters of serum half life around first dose on day of life 1 during hypothermia, and day of life 5 during normothermia
Change in Glutathione concentration in Basal ganglia | day of life 5
  GSH by MRS before, immediately after and up to 6h after NVD infusion on day of life 5

SECONDARY OUTCOMES:
Change in plasma oxidative stress markers | day 1 and 5
  isofurans measured by Liquid Chromatography-Mass Spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea Jenkins, MD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: Yes
after publication, upon request
Supporting Information: Study Protocol
Time Frame: after publication of main findings
Access Criteria: written request to PI

REFERENCES:
- [Background] Jenkins DD, Wiest DB, Mulvihill DM, Hlavacek AM, Majstoravich SJ, Brown TR, Taylor JJ, Buckley JR, Turner RP, Rollins LG, Bentzley JP, Hope KE, Barbour AB, Lowe DW, Martin RH, Chang EY. Fetal and Neonatal Effects of N-Acetylcysteine When Used for Neuroprotection in Maternal Chorioamnionitis. J Pediatr. 2016 Jan;168:67-76.e6. doi: 10.1016/j.jpeds.2015.09.076. Epub 2015 Nov 3. PMID 26545726
- [Background] Nie X, Lowe DW, Rollins LG, Bentzley J, Fraser JL, Martin R, Singh I, Jenkins D. Sex-specific effects of N-acetylcysteine in neonatal rats treated with hypothermia after severe hypoxia-ischemia. Neurosci Res. 2016 Jul;108:24-33. doi: 10.1016/j.neures.2016.01.008. Epub 2016 Feb 3. PMID 26851769
- [Background] Lowe DW, Fraser JL, Rollins LG, Bentzley J, Nie X, Martin R, Singh I, Jenkins D. Vitamin D improves functional outcomes in neonatal hypoxic ischemic male rats treated with N-acetylcysteine and hypothermia. Neuropharmacology. 2017 Sep 1;123:186-200. doi: 10.1016/j.neuropharm.2017.06.004. Epub 2017 Jun 6. PMID 28599922
- [Background] Lowe DW, Hollis BW, Wagner CL, Bass T, Kaufman DA, Horgan MJ, Givelichian LM, Sankaran K, Yager JY, Katikaneni LD, Wiest D, Jenkins D. Vitamin D insufficiency in neonatal hypoxic-ischemic encephalopathy. Pediatr Res. 2017 Jul;82(1):55-62. doi: 10.1038/pr.2017.13. Epub 2017 Jan 17. PMID 28099429
- [Background] Wiest DB, Chang E, Fanning D, Garner S, Cox T, Jenkins DD. Antenatal pharmacokinetics and placental transfer of N-acetylcysteine in chorioamnionitis for fetal neuroprotection. J Pediatr. 2014 Oct;165(4):672-7.e2. doi: 10.1016/j.jpeds.2014.06.044. Epub 2014 Jul 23. PMID 25064164
- [Result] Moss HG, Brown TR, Wiest DB, Jenkins DD. N-Acetylcysteine rapidly replenishes central nervous system glutathione measured via magnetic resonance spectroscopy in human neonates with hypoxic-ischemic encephalopathy. J Cereb Blood Flow Metab. 2018 Jun;38(6):950-958. doi: 10.1177/0271678X18765828. Epub 2018 Mar 21. PMID 29561203
- [Result] Sanchez-Illana A, Thayyil S, Montaldo P, Jenkins D, Quintas G, Oger C, Galano JM, Vigor C, Durand T, Vento M, Kuligowski J. Novel free-radical mediated lipid peroxidation biomarkers in newborn plasma. Anal Chim Acta. 2017 Dec 15;996:88-97. doi: 10.1016/j.aca.2017.09.026. Epub 2017 Sep 28. PMID 29137711